CLINICAL TRIAL: NCT03518203
Title: Early Intervention With Eculizumab to Treat Thrombotic Microangiopathy/Atypical Hemolytic Uremic Syndrome (TMA/aHUS)-Associated Multiple Organ Dysfunction Syndrome (MODS) in Hematopoietic Stem Cell Transplant (HCT) Recipients
Brief Title: Eculizumab to Treat Thrombotic Microangiopathy/Atypical Hemolytic Uremic Syndrome -Associated Multiple Organ Dysfunction Syndrome in Hematopoietic Stem Cell Transplant Recipients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-7119C
Record Dates: First submitted 2018-03-05; First posted 2018-05-08 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Thrombotic Microangiopathies; Atypical Hemolytic Uremic Syndrome; Multiple Organ Dysfunction Syndrome
Keywords: Hematopoietic Stem Cell Transplant
MeSH Terms: conditions — Thrombotic Microangiopathies; Atypical Hemolytic Uremic Syndrome; Multiple Organ Failure | interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Eculizumab (Experimental): All patients will receive eculizumab based on their weight for 24 weeks.
  Interventions: Drug: Eculizumab

INTERVENTIONS:
Drug: Eculizumab — Eculizumab will be administered as intravenous infusion (IV) over 60 minutes. The dosage form will be 300 mg single-use vials each containing 30 mL of 10 mg/mL sterile, preservative-free solution.
  Other Names: Soliris

SUMMARY:
Hematopoietic stem cell transplantation (HCT)-associated thrombotic microangiopathy (TMA) is an understudied complication of HCT that significantly affects transplant related morbidity and mortality. The investigators hypothesize that early intervention with complement blocker eculizumab will double survival in HCT recipients with high risk TMA, as compared to historical untreated controls. An optimal eculizumab dosing schedule can be determined for this population through eculizumab pharmacokinetic/pharmacodynamic (PK/PD) testing.

DETAILED DESCRIPTION:
This clinical trial is a prospective single arm multi-institution study in children and young adults undergoing allogeneic or autologous hematopoietic stem cell transplantation who will receive early therapy with eculizumab to prevent TMA-associated MODS after transplantation. The purpose of this research study is to examine efficacy of complement blocker eculizumab in HCT recipients with high risk TMA and to determine optimal eculizumab dosing regimen for HCT recipients with TMA using PK/PD studies. All patients will receive therapy based on their weight for 24 weeks. Survival will be assessed at 6 months from TMA diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any age undergoing allogeneic or autologous HCT
* Histologic TMA diagnosis OR clinical TMA diagnosis and presenting with high risk disease features including elevated plasma sC5b-9 above laboratory normal value (≥244ng/ml) and proteinuria measured as ≥30mg/dL of protein on random urinalysis x2 or protein/creatinine ratio ≥1mg/mg or patient receiving renal replacement therapy.
* Minimum weight of ≥ 5kg.

Exclusion Criteria:

* Known hypersensitivity to any constituent of the study medication.
* Subjects with unresolved serious Neisseria meningitides infection or progressive severe infection.
* Patients with diagnosis of TTP as defined by ADAMST13 activity test <10%.
* Patients previously treated with eculizumab or other complement blocker for TMA within the 60 days prior to first dose of study treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonata Jodele, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (3):
- United States (3):
  - Children's Hospital Los Angeles (CHLA), Los Angeles, California
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Jodele S, Dandoy CE, Aguayo-Hiraldo P, Lane A, Teusink-Cross A, Sabulski A, Mizuno K, Laskin BL, Freedman J, Davies SM. A prospective multi-institutional study of eculizumab to treat high-risk stem cell transplantation-associated TMA. Blood. 2024 Mar 21;143(12):1112-1123. doi: 10.1182/blood.2023022526. PMID 37946262

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Eculizumab
Started | 23
Completed | 21
Not Completed | 2
Not completed — The participant died on study prior to receiving 4 doses and was not evaluable. | 1
Not completed — Relapsed with primary malignancy within 6 months of TMA diagnosis making participant unevaluable. | 1

BASELINE CHARACTERISTICS:
Arm/Group | Eculizumab
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 17
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Survival
Description: Survival at 6 months after the date of TMA diagnosis
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 21
Participants | 15
Statistical Analysis 1: Comparison: Eculizumab; Test type: Equivalence — A binomial test was used to test 6 month survival in study cohort against an 18% historical rate; p < 0.0001, binomial test — The a priori threshold was 0.05; Proportion = 0.714

2. Secondary Outcome: Number of Participants With Organ Dysfunction
Description: Number of participants with organ dysfunction at 6 months after TMA diagnosis. Organ dysfunction definitions are listed in the protocol Appendix II that is uploaded to ClinicalTrials.gov site.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 15
Participants | 4

3. Secondary Outcome: Number of Participants With Organ Dysfunction
Description: Number of participants with organ dysfunction at 1 year after TMA diagnosis. Organ dysfunction definitions are listed in the protocol Appendix II that is uploaded to ClinicalTrials.gov site.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 13
Participants | 2

4. Secondary Outcome: Non-relapse Mortality
Description: Non-relapse mortality descriptively compared with historical controls at 1 year
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 21
Participants | 8

ADVERSE EVENTS:
Time Frame: Adverse Events were monitored from enrollment to 60 days after end of treatment, an average of 32 weeks. All-Cause Mortality was monitored up to 1 year.
Arm/Group | Eculizumab
All-Cause Mortality (participants affected / at risk) | 9/23
Serious Adverse Events (participants affected / at risk) | 19/23
Other Adverse Events (participants affected / at risk) | 22/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eculizumab (N=23)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Cardiac Tamponade (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2)
Decreased left ventricular ejection fraction (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Abdominal pain, right upper quadrant (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Fever (General disorders) | 3 (3)
Graft versus Host Disease (liver and gastrointestinal) (General disorders) | 1 (1)
Sinusoidal obstruction syndrome (Hepatobiliary disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Multi organ failure (Infections and infestations) | 3 (3)
Possible/Rule Out Sepsis (Infections and infestations) | 3 (3)
Sepsis (Infections and infestations) | 5 (5)
Platelet count decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Muscle weakness, lower limbs (Musculoskeletal and connective tissue disorders) | 1 (1)
Altered mental status (Nervous system disorders) | 2 (3)
Decreased level of consciousness (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Possible seizure (Nervous system disorders) | 1 (2)
Seizure (Nervous system disorders) | 3 (3)
Stroke (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 8 (8)
Renal failure (Renal and urinary disorders) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diffuse alveolar hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Worsening Hypoxia (due to diffuse alveolar damage) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary edema (related to fluid overload) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory decline (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 (10)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 3 (3)
Adenovirus infection (viral hepatitis) (Infections and infestations) | 1 (1)
Hemorrhagic shock, refractory (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eculizumab (N=23)
Anemia (Blood and lymphatic system disorders) | 2 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Increased cardiac troponin (Cardiac disorders) | 1 (1)
Biventricular dysfunction (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Ocular graft versus host disease (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
Graft versus host disease (Gastrointestinal disorders) | 2 (2)
Ileus (Gastrointestinal disorders) | 1 (1)
Lower GI hemorrhage (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Fever (General disorders) | 2 (4)
Generalized edema (General disorders) | 1 (1)
TMA reactivation unresponsive to treatment (General disorders) | 1 (1)
Adenoviremia (Infections and infestations) | 2 (2)
Bacteremia (Infections and infestations) | 4 (7)
BK viremia (Infections and infestations) | 1 (1)
Blood bilirubin increased (Infections and infestations) | 3 (3)
CMV viremia (Infections and infestations) | 1 (1)
CMV viremia reactivation (Infections and infestations) | 3 (3)
Endocarditis infective (Infections and infestations) | 1 (1)
Enterocolitis infections (Infections and infestations) | 1 (1)
Worsening enterocolitis (Infections and infestations) | 1 (1)
EBV reactivation (Infections and infestations) | 2 (2)
Fungal infection (right cheek, vaginal area) (Infections and infestations) | 1 (1)
Fungemia (Infections and infestations) | 2 (2)
Mucosal infection (eschar around nares) (Infections and infestations) | 1 (1)
Persistent C-Diff infection (Infections and infestations) | 1 (1)
Pulmonary, liver and splenic nodules, possible EBV (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Viral infection (HSV1 in blood and on skin) (Infections and infestations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Increased alanine aminotransferase (Investigations) | 8 (11)
Increased aspartate aminotransferase (Investigations) | 9 (10)
Neutrophil count decreased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 2 (2)
Renal tubular acidosis (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 14 (17)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness/pain trunk (left hip) (Musculoskeletal and connective tissue disorders) | 1 (1)
Worsened generalized muscle weakness (Nervous system disorders) | 1 (1)
Altered mental status (Nervous system disorders) | 1 (1)
Delirium (Nervous system disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1)
Vasovagal reaction (Nervous system disorders) | 1 (1)
End stage renal disease (or CKD) (Renal and urinary disorders) | 4 (4)
Hematuria (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tension pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin graft versus host disease (Skin and subcutaneous tissue disorders) | 2 (2)
Skin pain (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (3)
Hypotension (Vascular disorders) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1)
Disseminated adenovirus (Infections and infestations) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT03518203/Prot_SAP_001.pdf
  • Informed Consent Form (2020-08-31): https://cdn.clinicaltrials.gov/large-docs/03/NCT03518203/ICF_000.pdf